CLINICAL TRIAL: NCT01071824
Title: Prospective Randomised Study for Comparison of the Size of Limb of Transverse Coloplasty Pouch After Low Rectal Resection With Total Mesorectal Excision
Brief Title: Comparison of Limb Size of Transverse Coloplasty Pouch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Liestal (Other)
Responsible Party: Principal Investigator, Christoph A. Maurer, MD, Prof. Dr. med. Christoph A. Maurer, Kantonsspital Liestal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 303/08
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Colon Cancer
Keywords: size; limb; transverse coloplasty pouch; rectal resection; mesorectal excision; treatment outcome
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transverse coloplasty pouch (Short limb) (Active Comparator): The short limb is the standard technique of transverse coloplasty pouch.
  Interventions: Procedure: Transverse coloplasty pouch (Short limb)
- Transverse coloplasty pouch (Long limb) (Experimental): The long limb relates to straight coloanal anastomosis.
  Interventions: Procedure: Transverse coloplasty pouch (Long limb)

INTERVENTIONS:
Procedure: Transverse coloplasty pouch (Long limb) — Transverse coloplasty pouch with long limb
  Arms: Transverse coloplasty pouch (Long limb)
Procedure: Transverse coloplasty pouch (Short limb) — Transverse coloplasty pouch with short limb
  Arms: Transverse coloplasty pouch (Short limb)

SUMMARY:
The aim of the study is the comparison of pouch function with two different sizes of limb of transverse coloplasty pouch after rectal resection and total mesorectal excision.

DETAILED DESCRIPTION:
No detailed description necessary, see brief summary.

ELIGIBILITY:
Inclusion Criteria:

* all patients in need of rectal resection due to benign or malign disease
* >=18 years

Exclusion Criteria:

* anamnestic rectal resection
* life expectancy of less than 2 years
* pregnancy
* <18 years
* missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2009-06; Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pouch function 4 month after closure of protective ileostomy. | 4 month

SECONDARY OUTCOMES:
Pouch function 2 and 12 month respectively after closure of protective ileostomy. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Maurer, Prof, Principal Investigator — Kantonsspital Liestal
Locations (1):
- KS Liestal, Liestal, Basel-Landschaft, Switzerland